CLINICAL TRIAL: NCT00986635
Title: Effect of Rivaroxaban on Coagulation Parameters- an ex Vivo Study
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Prof. Dr. Edelgard Lindhoff-Last, MD, Vascular Medicine, Johann Wolfgang Goethe University Hospital Frankfurt/Main
Other Study IDs: RIV139/09
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2009-09

CONDITIONS: Differences in Laboratory Coagulation Parameters
Keywords: Activated partial thromboplastin time; Thrombin clotting Time; Anti-Xa-activity; Factor X-activity; Factor XIII-activity; Antithrombin (based on factor II); Antithrombin (based on factor X<9

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Plasma samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Rivaroxaban represent a new class of anticoagulation agents. As an oral direct factor Xa inhibitor it has been effective in preventing venous thromboembolism in patients undergoing elective orthopaedic surgery. This ex vivo study is undertaken to investigate the ex-vivo effects of Xarelto® on different coagulation parameters.

DETAILED DESCRIPTION:
To validate the effects of Rivaroxaban on coagulation parameters plasma samples of patients after hip or knee replacement surgery treated with Rivaroxaban 10 mg/d are investigated.

Plasma samples are obtained by blood collection before, after 2 hours and after 12 hours after Rivaroxaban dosing in steady state (on 3rd - 5th day).

Several techniques, including clot-based tests, chromogenic assays and ELISA´s are used for coagulation assays in our coagulation laboratory Frankfurt/Main. The influence of Rivaroxaban on different coagulation assays should be investigated in our coagulation laboratory.

ELIGIBILITY:
Inclusion Criteria:

* patients after hip or knee replacement surgery treated with Rivaroxaban 10 mg/d
* must be able to accept blood sampling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients after hip or knee replacement surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Mani, PhD, Principal Investigator — Johann Wolfgang Goethe University Hospital Frankfurt/Main Germany
Locations (1):
- University Hospital Frankfurt, Frankfurt am Main, Germany

REFERENCES:
- [Derived] Mani H, Hesse C, Stratmann G, Lindhoff-Last E. Ex vivo effects of low-dose rivaroxaban on specific coagulation assays and coagulation factor activities in patients under real life conditions. Thromb Haemost. 2013 Jan;109(1):127-36. doi: 10.1160/TH12-04-0228. Epub 2012 Nov 8. PMID 23138190